CLINICAL TRIAL: NCT03463980
Title: Compassion Meditation and ReliefLink App for Suicidal, Low-Income, African Americans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated during the pandemic as data collection could not be completed any further, and personnel changes did not allow for completion. At the time of termination, enough data was collected for a publication, all benchmarks were met.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nadine Kaslow, PhD, Professor & Chief Psychologist, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00038057
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Suicidal Ideation
Keywords: Meditation; African American; Randomized controlled trial
MeSH Terms: conditions — Suicidal Ideation | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compassion meditation (CM) (Experimental): The CM participants will attend six weekly sessions (each 120 minute), and will be video and/or audiotaped. Each weekly CM session will entail a 30 minute check-in regarding the participants' levels of suicidal ideation, as well as a discussion of current life stress and weekly meditation practice; a 30 minute didactic session that will describe the meditative technique introduced during the week; and a 30 minute guided meditation session. Participants will be encouraged to meditate at least 30 minutes a day and will be asked to track their daily meditation time and bring in their tracking sheet to each session.
  Interventions: Behavioral: Compassion meditation (CM)
- Support group (SG) (Active Comparator): SG participants will attend six weekly sessions, 90 minutes in length. It will be unstructured. Participants will use this time to talk about current concerns and to receive support and guidance from other group members and the leaders.
  Interventions: Behavioral: Support group (SG)

INTERVENTIONS:
Behavioral: Compassion meditation (CM) — CM session: 30 minute check-in regarding the participants' levels of suicidal ideation, as well as a discussion of current life stress and weekly meditation practice; a 30 minute didactic session that will describe the meditative technique introduced during the week; and a 30 minute guided meditation session. Participants are also encouraged to meditate at least 30 minutes a day.
  Arms: Compassion meditation (CM)
Behavioral: Support group (SG) — SG session: 90 minutes to talk about current concerns and to receive support and guidance from other group members and the leaders.
  Arms: Support group (SG)

SUMMARY:
The purpose of this study is to conduct a pilot randomized controlled trial (RCT) with low-income, suicidal African American women and men that compares the relative effectiveness of compassion meditation (CM) versus a support group (SG) .

DETAILED DESCRIPTION:
The purpose of this study is to conduct a pilot randomized controlled trial (RCT) with low-income, suicidal African American women and men that compares the relative effectiveness of compassion meditation (CM) versus a support group (SG) for (1) reducing psychological distress (suicidal ideation, depressive symptoms, and shame); (2) bolstering interpersonal connectedness; and (3) enhancing self-compassion and mindfulness. It is hypothesized that at post-intervention and follow-up, compared to individuals in the SG, those in the CM intervention will endorse less psychological distress (suicidal ideation, depressive symptoms, and shame), more interpersonal connectedness, and greater levels of self-compassion and mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as African American or Black
* speak English
* present to medical and psychiatric emergency rooms at Grady Health System following a suicide attempt
* moderate level of intent associated with the attempt (SSI >= 8 required)
* Mini Mental State Exam (MMSE) score > 22

Exclusion Criteria:

* significant cognitive impairments (MMSE < 22)
* active psychosis (diagnosed based on Psychotic Screen (PS))
* imminently life-threatening medical condition

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 456 (Actual)
Dates: Start 2010-05-13 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Change in Beck Scale for Suicide Ideation (BSS) score | Pre-intervention - baseline (T1), post-intervention - at completion of 6 weekly sessions (T2), and at 6 week follow-up (T3)
  The BSS is a self-report 19-item scale preceded by five screening items. The BSS and its screening items are intended to assess a patient's thoughts, plans and intent to commit suicide. All 24 items are rated on a three-point scale (0 to 2) total scores could range from 0 to 48. No specific cut-off scores exist to classify severity or guide patient management. Increasing scores reflect greater suicide risk, and any positive response merits investigation.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory II (BDI-II) score | Pre-intervention - baseline (T1), post-intervention - at completion of 6 weekly sessions (T2), and at 6 week follow-up (T3)
  The BDI is a self-report 21-item scale used to assess the current severity of depression. Each item is rated on a four-point scale (0 to 3) with possible total scores ranging from 0 to 63. Scores provide a measure of the severity of self-reported depression: 0 -9 minimal, 10 -16 mild, 17-29 moderate, and 30 - 63 severe.
Change in Experience of Shame Scale (ESS) score | Pre-intervention - baseline (T1), post-intervention - at completion of 6 weekly sessions (T2), and at 6 week follow-up (T3)
  The Experiences of Shame Scale (ESS) is a 25 item inventory that measures the experience of shame about a variety of areas including shame about one's body, personal habits, manner with others, personal ability, whether one has said or done something wrong (e.g. "Have you felt ashamed of any of your personal habits?") over the past month.. Participants are asked to answer questions on a 4 point Likert scale from "not at all" to "very much."
Change in Levels of Self-Criticism Scale (LOSC) score | Pre-intervention - baseline (T1), post-intervention - at completion of 6 weekly sessions (T2), and at 6 week follow-up (T3)
  The Levels of Self-Criticism Scale (LOSC), which has 22 items assessing comparative self-criticism and internalized self-criticism, will be used to measure the level of self-criticism. The LOSC measures both comparative self-criticism (e.g. "I fear that if people get to know me too well, they will not respect me.") and internalized self-criticism (e.g. "Failure is a very painful experience for me."). Participants are asked to rate each item on a 7 point Likert scale from "not at all" to "very well."
Change in Social Support Behaviors Scale (SSB) score | Pre-intervention - baseline (T1), post-intervention - at completion of 6 weekly sessions (T2), and at 6 week follow-up (T3)
  is interpersonal connectedness. It will be evaluated using the 45 item Social Support Behaviors Scale (SSB), which includes five modes of social support separately for family and friends and these subscale have been confirmed with a multi-ethnic sample. Respondents rate, on a scale of 1 to 5: 1- no one would provide the support, to 5 - most (family/friends) would do this.
Change in Self-Compassion Scale (SCS) score | Pre-intervention - baseline (T1), post-intervention - at completion of 6 weekly sessions (T2), and at 6 week follow-up (T3)
  particularly relevant to the focus of the intervention, namely self-compassion and mindfulness. The 26-item Self-Compassion Scale (SCS) includes six domains of self-compassion: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identified. Scores on the SCS are correlated with lower levels of depression and anxiety and better life satisfaction.
Change in Five Facet Mindfulness Questionnaire (FFMQ) score | Pre-intervention - baseline (T1), post-intervention - at completion of 6 weekly sessions (T2), and at 6 week follow-up (T3)
  The Five Facet Mindfulness Questionnaire (FFMQ) will be used to assess five elements of mindfulness, observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. The measure includes 39-items that are rated on a 1 to 5 point Likert-type scale assessing five facets.
Change in Behavior Monitoring Form (BMF) score | Weekly during participation in the study up to 3 months
  The Behavior Monitoring Form (BMF) assesses suicidal behavior (levels of hopelessness, depressive feelings, stress, suicidal thoughts, suicidal actions) in the prior week; items are rated on a 5 point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Kaslow, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Health System (non-CRN), Atlanta, Georgia, United States

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832